CLINICAL TRIAL: NCT04565769
Title: Cognitive Function in Patients Treated for Melanoma With Adjuvant Immune Checkpoint Inhibitors: A Controlled Prospective Observational Study
Brief Title: Cognitive Function in Melanoma Patients Treated With Adjuvant Immune Checkpoint Inhibitors
Status: Active, not recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Josefine Tingdal Taube, Cand.psych., Ph.d.-fellow, Aarhus University Hospital
Other Study IDs: 2016-051-000001-1730
Record Dates: First submitted 2020-09-16; First posted 2020-09-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Melanoma; Cognitive Impairment; Fatigue; Sleep; Depression, Anxiety; Quality of Life; Inflammation; Sickness Behavior; Cancer-related Cognitive Impairment
Keywords: Immune Checkpoint Inhibitors; Melanoma; Cancer-related Symptoms; Cognitive Dysfunction
MeSH Terms: conditions — Melanoma; Cognitive Dysfunction; Fatigue; Depression; Anxiety Disorders; Inflammation; Illness Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer patients with melanoma: Forty seven cancer patients with melanoma included prior to treatment with ICI.
- Healthy controls: Fifthy three age- and gender- matched healthy controls.

SUMMARY:
Immune checkpoint inhibitors (ICIs) are a group of novel immunotherapies that boost the body's own defense against the cancer by improving the immune system's ability to recognize and destroy cancer cells. While it is relatively well-documented that conventional cancer treatments (e.g., chemotherapy) are associated with cognitive impairment, virtually nothing is yet known about effects on cognition during and after ICI treatment. Due to significantly improved survival rates after ICI treatments, it becomes important to map possible adverse effects associated with these treatments. The investigators therefore investigate possible changes in cognitive function in a group of cancer patients from prior to ICI treatment to nine months later. A gender- and age- matched healthy control group will serve as a comparison. The study has the potential to broaden our understanding of associations between cognition, the brain, and the immune system and to provide clinically relevant knowledge about possible cognitive impairments associated with immunotherapy.

DETAILED DESCRIPTION:
This controlled prospective observational study will include two groups with a total of 84 participants. A total of 42 patients diagnosed with melanoma, referred to treatment with ICI will be enrolled in the study and examined prior to treatment with ICI (baseline), at eight weeks following baseline (T2), at 24 weeks following baseline (T3) and 12 weeks after treatment completed (T4). A total of 42 gender- and age- matched healthy controls will be included and assessed at similar time points. Assessments will include a battery of neuropsychological tests, questionnaires, blood samples, and Magnetic Resonance Imaging (MRI).

The main objectives of the study are to investigate:

1. Changes in cognitive functions over the course of treatment with ICIs.
2. Possible associations between changes in cognitive function and immune markers during and following ICI treatment.
3. Possible associations between changes in cognitive function and changes in brain morphology.
4. Changes over time in other possible adverse effects of ICI treatment, including psychological distress, sleep disturbances, and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of melanoma and scheduled for ICI treatment at Aarhus University Hospital (AUH), Denmark. The healthy control group will consist of an age- and gender- matched sample of participants.

Exclusion Criteria:

* Previous treatment with immunotherapy
* Neurodegenerative diseases (dementia etc.)
* Substance abuse
* Known progressive psychiatric diseases (e.g., Schizophrenia)
* Other confirmed diagnoses with underlying cognitive impairment
* Insufficient Danish proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with melanoma and scheduled for ICI treatment at Aarhus University Hospital, Denmark. Controls will be healthy volunteers of cancer-free participants matched on age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Attention | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in attention as measured with WAIS-IV The Digit Span Forwards (scores with a minimum of 0 points to a maximum of 16 points - higher scores mean a better outcome)
Attention | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in attention as measured with Paced Auditory Serial Addition Test (scores ranging from a minimum of 0 and a maximum of 60 with higher scores indicating a better outcome)
Processing Speed | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in processing speed as measured with WAIS-IV The Digit Symbol coding (scores ranging from a minimum of 0 and a maximum of 135 with higher scores indicating a better outcome)
Processing Speed | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in processing speed as measured with Trail Making Test A (outcome is time in seconds)
Working memory | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in working memory as measured with WAIS-IV The Digit Span Backwards (scores with a minimum of 0 points to a maximum of 16 points - higher scores mean a better outcome)
Working memory | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in working memory as measured with WAIS-IV The Digit Span Ranking (scores with a minimum of 0 points to a maximum of 16 points - higher scores mean a better outcome)
Learning and memory | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in learning and memory as measured with the Hopkins Verbal Learning Test - Revised (part 1 include a minimum score of 0 and a maximum score of 36 with higher score indicating a better outcome, part 2 include a minimum score of 0 and a maximum score of 12 with higher scores indicating better outcomes)
Learning and memory | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in learning and memory as measured with Brief Visuospatial Memory Test - Revised (part 1 include a minimum score of 0 and a maximum score of 18 with a higher score indicating a better outcome, part 2 include a minimum score of 0 and a maximum score of 6 with higher scores indicating better outcomes)
Visuospatial ability | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in visuospatial ability as measured with WAIS-IV Matrix Reasoning (scores with a minimum of 0 and a maximum of 26 with higher scores indicating better outcomes)
Verbal fluency | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in verbal fluency as measured with the Controlled Oral Word Association Test, letter and animal (as many words as possible, more words indicating a better outcome. No maximum value)
Executive function | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in executive function as measured with the Trail Making Test B (outcome is time in seconds)

SECONDARY OUTCOMES:
Cancer-related fatigue | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in fatigue severity as measured with The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT fatigue) scale (range from 0 to 52. Items are reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatigue)
Sleep quality | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in sleep quality as measured with the Insomnia Severity Index (ISI) (scores ranging from a minimum of 0 and a maximum of 28 with higher scores indicating higher levels of insomnia)
Sleep quality | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in sleep quality as measured with the Pittsburgh Sleep Quality Index (PSQI) (scores ranging form a minimum of 0 indicating no difficulty and a maximum of 21 indicating severe difficulties in all areas related to sleep)
Perceived cognitive functioning | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in perceived cognitive functioning as measured with The Patient Assessment of Own Functioning Inventory (PAOFI) (outcome is scores ranging from a minimum of 35 to a maximum of 210)
Depression/Anxiety | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in depression/anxiety as measured with the Hospital Anxiety and Depression Scale (HADS) (range from a minimum score of 0 to a maximum score of 21 in which a higher scores mean higher levels of depression/anxiety)
Sickness behavior | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in subjective sickness behavior as measured with the Sickness Questionnaire (SicknessQ) (scores ranging from a minimum of 0 and a maximum of 30 with higher scores indicating worse outcome)
Health-related quality of life | Baseline, and week 8, 24 and 12 weeks after completed treatment
  Changes in health-related quality of life as measured with The European Organization for Research and Treatment of Cancer, Quality of Life questionnaire for cancer patients (EORTC QLQ-C30) (all of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.)
Moderator: genotype | Baseline
  Genotype of COMT and APOE4
  Genotype of COMT
Inflammatory immune markers | Baseline, and week 8, 24 and 12 weeks after completed treatment
  TNF-α, IL-6, IL-8, IL-21, CRP, IP-10 and MCP-1 extracted from blood samples
Brain grey matter | Baseline and week 24.
  Changes in brain grey matter as measured with T1-weighted MRI
Brain white matter | Baseline and week 24.
  Changes in brain white matter as measured with T1-weighted MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided